CLINICAL TRIAL: NCT01609244
Title: Bilevel Versus Servoventilation in Complex Sleep Apnea
Acronym: CSA-FKKG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Kloster Grafschaft (Other)
Responsible Party: Principal Investigator, Dominic Dellweg, M.D., Attending physician sleep laboratoy and home mechanical ventilation unit, Krankenhaus Kloster Grafschaft
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA-2010
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Complex Sleep Apnea; CPAP Induced Central Sleep Apnea
Keywords: Sleep apnea; central sleep apnea; bilevel; servoventilation; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilevel (Active Comparator): Bilevel therapy
  Interventions: Device: Bilevel therapy (somnovent ST 22, Weinmann, Hamburg, Germany)
- Servoventilation (Active Comparator): servoventilation therapy
  Interventions: Device: servoventilation (Somnovent CR, Weinmann, Hamburg, Germany)

INTERVENTIONS:
Device: Bilevel therapy (somnovent ST 22, Weinmann, Hamburg, Germany) — nighttime positive airway therapy for 6 weeks
  Arms: Bilevel
Device: servoventilation (Somnovent CR, Weinmann, Hamburg, Germany) — nighttime positive airway therapy for 6 weeks
  Arms: Servoventilation

SUMMARY:
Randomized trial to evaluate the performance of Bilevel vs. Servoventilation in patients with complex sleep apnea during continuous positive airway pressure (CPAP) treatment.

DETAILED DESCRIPTION:
Patients with primary obstructive sleep apnea, who develop complex sleep apnea after CPAP treatment of 4-6 weeks duration were randomized to either receive Bilevel of Servoventilation treatment. Parameters of sleep as well as apnea-hypopnea indices are to be compared.

ELIGIBILITY:
Inclusion Criteria:

Predominant obstructive apnea without treatment Predominant central apnea with CPAP treatment

Exclusion Criteria:

primary central sleep apnea non-compliance to CPAP therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | at 6 weeks
  apneas and hypopneas under therapy

SECONDARY OUTCOMES:
Percentage slow wave sleep, percentage rapid eye movement (REM) sleep, Arousal index, sleep time, sleep efficacy | at 6 weeks
  parameters of sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dellweg, MD, Study Chair — FKKG
Locations (1):
- Kloster Grafschaft, Schmallenberg, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Kuzniar TJ, Pusalavidyasagar S, Gay PC, Morgenthaler TI. Natural course of complex sleep apnea--a retrospective study. Sleep Breath. 2008 May;12(2):135-9. doi: 10.1007/s11325-007-0140-z. PMID 17874254
- [Derived] Dellweg D, Kerl J, Hoehn E, Wenzel M, Koehler D. Randomized controlled trial of noninvasive positive pressure ventilation (NPPV) versus servoventilation in patients with CPAP-induced central sleep apnea (complex sleep apnea). Sleep. 2013 Aug 1;36(8):1163-71. doi: 10.5665/sleep.2878. PMID 23904676